CLINICAL TRIAL: NCT04158284
Title: KRANIOPHARYNGEOM Registry 2019 Multicenter Registry for Patients With Childhood-onset Craniopharyngioma, Xanthogranuloma, Cysts of Rathke's Pouch, Meningioma, Pituitary Adenoma, Arachnoid Cysts
Brief Title: Multicenter Registry for Patients With Childhood.Onset Craniopharyngioma, Xanthogranuloma, Cysts of Rathke's Pouch, Meningioma, Pituitary Adenoma, Arachnoid Cysts
Status: Recruiting | Type: Observational
Sponsor: Klinikum Oldenburg gGmbH (Other)
Collaborators: German Society for Pediatric Oncology and Hematology GPOH gGmbH (Other); Deutsche Gesellschaft für Kinderendokrinologie und Diabetologie (DGKED) (Unknown); Deutsche Gesellschaft für Endokrinologie (DGE) (Unknown); Arbeitsgemeinschaft Pädiatrische Radioonkologie (APRO) (Unknown); Deutschen Gesellschaft für Radioonkologie (DEGRO) (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. med. Hermann Mueller, Professor MD, Klinikum Oldenburg gGmbH
Other Study IDs: KRANIOPHARYNGEOM Registry 2019
Record Dates: First submitted 2019-10-10; First posted 2019-11-08 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Craniopharyngioma; Obesity
Keywords: Quality of life; Endocrinology; Oncology; Hypothalamus; Irradiation; Neurosurgery; Pediatric Brain tumors
MeSH Terms: conditions — Craniopharyngioma; Obesity; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
KRANIOPHARYNGEOM Registry 2019 will prospectively collect and descriptively analyse data on diagnostics, treatment, and follow-up of patients with craniopharyngioma. In continuation of preceding studies also patients with xanthogranuloma, meningioma, pituitary adenoma, prolactinoma and cystic intracranial malformations will be registered.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with craniopharyngioma for the first time
2. Age at diagnosis 18 years or less of age
3. Agreement from patient's parents or legal guardian as well as the patient

Exclusion Criteria:

1. Age at diagnosis over 18 years of age
2. Diagnosis different from craniopharyngioma

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Newly diagnosed patients (≤ 18 years of age) with childhood-onset craniopharyngioma
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 3 years follow-up
  Overall survival as measured by Kaplan Meyer analyses
Progression-free Survival (PFS) | 3 years follow-up
  Progression-free survival as measured by Kaplan Meyer analyses

SECONDARY OUTCOMES:
Quality of life (QoL) | 3 years follow-up
  Domains of the PedQol instrument (questionnaire for assessment of health-related QoL in childhood cancer patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Oldenburg, Oldenburg, Lower Saxony, Germany

REFERENCES:
- [Derived] Sowithayasakul P, Beckhaus J, Ozyurt J, Bison B, Friedrich C, Muller HL. Prolactin serum concentrations in childhood-onset craniopharyngioma patients. J Endocrinol Invest. 2025 Sep;48(9):2041-2051. doi: 10.1007/s40618-025-02622-4. Epub 2025 Jun 7. PMID 40481916
- [Derived] Mann-Markutzyk LV, Beckhaus J, Ozyurt J, Mehren A, Friedrich C, Muller HL. Daytime sleepiness and health-related quality of life in patients with childhood-onset craniopharyngioma. Sci Rep. 2025 Mar 19;15(1):9407. doi: 10.1038/s41598-025-94384-5. PMID 40108339
- [Derived] Wagener K, Beckhaus J, Boekhoff S, Friedrich C, Muller HL. Sporadic and neurofibromatosis type 2-associated meningioma in children and adolescents. J Neurooncol. 2023 Jul;163(3):555-563. doi: 10.1007/s11060-023-04344-0. Epub 2023 Jul 4. PMID 37402092
- [Derived] Beckhaus J, Friedrich C, Boekhoff S, Calaminus G, Bison B, Eveslage M, Timmermann B, Flitsch J, Muller HL. Outcome after pediatric craniopharyngioma: the role of age at diagnosis and hypothalamic damage. Eur J Endocrinol. 2023 Mar 2;188(3):lvad027. doi: 10.1093/ejendo/lvad027. PMID 36857103